CLINICAL TRIAL: NCT05578183
Title: Therapeutic Efficacy and Mechanism of Personalized Theta Burst Stimulation on Working Memory Impairment in Patients After Stroke
Brief Title: Therapeutic Effect of Transcranial Magnetic Stimulation on Memory Impairment in Patients After Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been registed in ChiCTR and apply for withdrawing.
Sponsor: China Rehabilitation Research Center (Other Government)
Responsible Party: Principal Investigator, Hao Zhang, Professor, China Rehabilitation Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZhang
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Stroke Sequelae; Cognitive Impairment
Keywords: stroke; cognitive impairment; transcranial magnetic stimulation; Functional Magnetic Resonance Imaging; event related potential
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- high dose TBS group (Experimental): parameters: pattern: intermittent TBS (iTBS; 2 seconds of TBS are delivered every 10 seconds), TBS consists of pulses applied in bursts of 3 at 50 Hz with an interburst interval at 5 Hz
  Interventions: Device: theta burst stimulation
- low dose TBS group (Experimental): parameters: pattern: intermittent TBS (iTBS; 2 seconds of TBS are delivered every 10 seconds), TBS consists of pulses applied in bursts of 3 at 50 Hz with an interburst interval at 5 Hz
  Interventions: Device: theta burst stimulation
- high dose sham TBS group (Sham Comparator): parameters: pattern: intermittent TBS (iTBS; 2 seconds of TBS are delivered every 10 seconds), TBS consists of pulses applied in bursts of 3 at 50 Hz with an interburst interval at 5 Hz
  Interventions: Device: sham stimulation
- low dose sham TBS group (Sham Comparator): parameters: pattern: intermittent TBS (iTBS; 2 seconds of TBS are delivered every 10 seconds), TBS consists of pulses applied in bursts of 3 at 50 Hz with an interburst interval at 5 Hz
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: theta burst stimulation — expect for the TBS, all patients get cognitive training alike on a training system in medical center.
  Other Names: Cognitive training
  Arms: high dose TBS group; low dose TBS group
Device: sham stimulation — expect for the TBS, all patients get cognitive training alike on a training system in medical center.
  Other Names: Cognitive training
  Arms: high dose sham TBS group; low dose sham TBS group

SUMMARY:
The goal of this clinical trial is to test the therapeutic effect of theta burst stimulation (TBS), which is one of stimulus pattern of repetitive transcranial magnetic stimulation, in patients with post stroke cognition impairment (PSCI). The main questions it aims to answer are:

1. To explore the therapeutic effect of TBS to patients with PSCI.
2. To compare effect of TBS with different dose.
3. To explore the mechanism of TBS by functional magnetic resonance imaging (fMRI).

Participants will be asked to do:

1. Treated with TBS and cognitive training for 3 weeks (15 days).
2. Assessed with several scales, including Mini-mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Loewenstein Occupational Therapy Cognitive Assessment (LOTCA), Wechsler Adult Intelligence Scale-revised in China (WAIS-RC), Wechsler Memory Scale (WMS) before and after treatment.
3. Perform the resting fMRI, electroencephalogram (EEG) and event related potential before and after treatment.

Researchers will compare high-dose group, low-dose group and sham group to see if TBS play a role in PSCI and if the effect of high dose TBS was stronger than low dose.

DETAILED DESCRIPTION:
the procedure of study

1. Patients were recruited and agreed with Informed Consent.
2. All patients were assessed with MMSE, MoCA, LOTCA, WAIS and WMS, meanwhile they conduct fMRI and EEG. Target of TBS set at dorsolateral prefrontal cortex (DLPFC).
3. TBS was performed for 15 days (5 days * 3 weeks).
4. Within 3 days after TBS, all patients were assessed with MMSE, MoCA, LOTCA, WAIS and WMS, meanwhile they conduct fMRI and EEG.
5. Data acquisition and analysis.

ELIGIBILITY:
Inclusion Criteria:

* First-time stroke patients, meeting the diagnostic criteria set by the Fourth National Conference of Cerebrovascular Diseases in 1995, and the course of stroke
* range from 1 to 12 months;
* The vital signs are stable and no progress in neurological signs;
* Education level: Primary school or above, and meeting one of the following conditions: MMSE scale ≥ 10 points, and indicating memory decline, with digit span or delayed memory defects.
* Patients or their family members sign the informed consent form.

Exclusion Criteria:

* Contraindications or high risks for TBS, such as epilepsy, intracranial metal implants, skull repair;
* Contraindications for fMRI, such as metal implants or claustrophobia; refuse fMRI;
* drug/alcohol dependence;
* Cognition or memory dysfunction before the onset;
* Patients who refuse to cooperate, or can't complete cognitive assessment due to other reasons, such as visual and auditory disturbance, aphasia, agnosia, apraxia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Montreal Cognitive Assessment scale | 1. finished in 3 days before TBS stimulation. 2. finished in 3 days after stimulation.
  one of the most used scales to assess cognition and screen person with cognitive impairment in the world. The minimum and maximum values range from 0 to 30. Higher score means better cognition level.

SECONDARY OUTCOMES:
Change from Baseline Mini-mental State Examination scale | 1. finished in 3 days before TBS stimulation. 2. finished in 3 days after stimulation.
  Easy to use and one of the most used scales to screen person with cognitive impairment in the world. The minimum and maximum values range from 0 to 30. Higher score means better cognition level.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhang, Study Director — China Rehabilitation Research Center
Locations (1):
- China rehabilitation research center, Beijing, Beijing Municipality, China